CLINICAL TRIAL: NCT04487964
Title: Evaluation of The Potential Therapeutic Effects of Licorice and Boswellia Serrata Gum in Egyptian Patients With COVID-19 as a Complementary Medicine
Brief Title: Complementary Intervention for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Adel Gomaa, Professor of medical pharmacology, Egyptian Biomedical Research Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0925-0586
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Glycyrrhiza glabra extract; Frankincense

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the conventional therapy according to the MOH protocol. (Active Comparator): Patients who are receiving conventional therapy according to the MOH protocol.
  Interventions: Dietary Supplement: Licorice extract
- conventional therapy +Liquorice cap and Boswellia Serrata gum (Active Comparator): Patients will receive Liquorice cap and Boswellia Serrata gum in addition to conventional therapy
  Interventions: Dietary Supplement: Licorice extract

INTERVENTIONS:
Dietary Supplement: Licorice extract — LICORICE CAPSULES; 250 mg standardized extract (25% Glycyrrhizin - 62.5 mg) For 10 days, with measuring blood pressure daily.
  Dose:
  One capsule, twice daily, before meals. Boswellia serrata Gum Resin; B. serrate contains volatile oils (5-15%), pure resin (55-66%), and mucus (12-23%). The resin contains terpenoids, phenolic compounds, flavonoids, and phenylpropanoids. More than 12 different Boswellic acids have been identified, the amounts of 11-keto-β-boswellic acid KBA is 3-4.7% and acetyl-11-keto-β-boswellic acid(AKBA) is 2.2-2.9%, Dose: 2 gm, 4 times daily For 15 days, Boswellia Gum Resin is administered by chewing for a half-hour
  Other Names: Boswellia serrata Gum

SUMMARY:
Boswellia Serrata gum and Licorice extract are two nutritional agents that have pharmacological actions that could support the medical intervention for COVID-19. They have broad antiviral activity, anti-inflammatory, anti-lung injury, antibacterial activity, antithrombic formation, and immunomodulatory activity.

The study will be conducted after January 18, 2017

DETAILED DESCRIPTION:
Since last December 2019, a syndrome of severe pneumonia associated with the coronavirus disease 2019 (COVID-19) emerged in Wuhan, Hubei Province, China. It is highly contagious and rapidly spread to many other parts of China and almost all countries all over the world, representing one of the most aggressive pandemics ever reported.

To date, April 21, 2020, More than 2.5 million persons were infected and more than 171.000 deaths with more fears all over the world from the multiplication of the total deaths. This huge no. of patients made a horrible pressure on health care facilities in all countries and lots of patients were not able to receive the appropriate medical care in hospitals WHO declared that to date, there is no specific medicine recommended to prevent or treat the novel coronavirus. However, in China, historically, when the outbreak started, Traditional Chinese medicine (TCM) approaches including oral administration of preventive herbal formulae, wearing TCM sachets, indoor herbal medicine fumigation, etc. were recommended for prevention and treatment.

For example, in 2003, TCM approaches were used to prevent and treat severe acute respiratory syndrome (SARS) which was the most serious infectious disease outbreak in China prior to the COVID-19. In 2009, during the pandemic of H1N1 influenza around the world, the National Administration of Traditional Chinese Medicine of China issued a CM prevention program, which included 4 Chinese herbal medicine (CHM) formulae for adults of different CM body constitutions and one for children. The current outbreak of COVID-19 resulted in many provinces in China issuing CM prevention and control programs, among which the prevention programs are mainly oral CHM formulae.

Glycyrrhizin, a component of many formulae, has reported having anti-inflammatory, antiviral and antioxidant properties. Also, Boswellia Gum Resin has many active components that have many medicinal properties such as antimicrobial, antioxidant, antifungal, anti-inflammatory, immuno-modulatory.

Efficacy:

1. The two agents have broad-spectrum antiviral effects in-vitro and in in-vivo in preclinical and clinical studies:

   A. There are clinical studies about the efficacy of licorice in severe acute respiratory syndrome-related coronavirus, This can be of major importance in the coronavirus infections, since immunodeficiency patients may be particularly at risk.

   B. There are traditional use and clinical experience of Chinese traditional Medicine containing licorice in the treatment of COVID 19.
2. The two agents have anti-inflammatory effects and blocking the production of cytokines which are the main causes for the severity of diseases.
3. The two agents have antioxidant effects, prevent tissue damages in the lungs.
4. The two agents inhibit the airway mass hyperplasia so, they alleviate anoxia state and improve clinical symptoms.
5. The two agents are used in the treatment of bronchial asthma and respiratory inflammatory disorders.
6. Licorice has antithrombin and antiplatelet effects so, it alleviates the hypercoagulation induced by COVID 19.
7. Licorice enhances the production of interferon-gamma that has high activity against the replication of the virus.

Safety:

1. Licorice and Boswellia Gum Resin had been considered as a food supplement or nutritional agents, so they have high safety margins in recommended doses, However, there is a contraindication for the use of licorice in non controlled hypertensive patients.
2. Hypertensive patients and patients sensitive to hypokalemia are excluded from this study. Regarding other patients, many studies documented that Hypertension may develop as an adverse reaction after chronic use of large doses.
3. Excessive consumption of licorice for a long time (more than 2 mg/kg/day of pure glycyrrhizinic acid, a licorice component) may result in adverse effects, such as hypokalemia, increased blood pressure, and muscle weakness. People with previously existing heart or kidney problems may be more susceptible to GZA and licorice poisoning. It is important to monitor the amount of licorice consumed in order to prevent toxicity.

More interesting, It has been shown that monoammonium glycyrrhizinate injection or glycyrrhizic acid exerts a protective influence on myocardial ischemic injury induced by isoproterenol by inhibiting oxidative stress and regulating Ca2+ homeostasis, therefore, it may be useful in the management of myocardial ischemic injury.

Isoliquiritigenin has reported having a significant anti-platelet action in vivo by inhibiting cyclooxygenase and lipoxygenase or peroxidase activity in platelets.

Glycyrrhizin (GL) elicits effective antithrombotic action (prevent thrombosis), as it was considered as an effective thrombin inhibitor.

However, the most important side effect is the induction of hypertension, and it can induce what appears to be pseudohyperaldosteronism, due to glycyrrhetinic acid the main active component of the root. Glycyrrhetinic acid and metabolites block the 11 beta-hydroxysteroid dehydrogenase type 2 and also bind mineralocorticoid receptors directly, acting as agonists.

Boswellia serrate (B.serrata) is used traditionally to treat chronic inflammatory diseases such as in acute systemic inflammation, accompanied liver dysfunction, and chronic inflammatory diseases. Recent studies show that Boswellia serrate can improve the clinical outcomes along with conventional therapies in ischaemic stroke. This action is due to the anti-inflammatory properties of the main bioactive compounds Boswellic acids (BAs). It inhibits the pro-inflammatory cytokines such as interleukin-1 β (IL-1 β), tumor necrosis factor-α (TNF-α), interferon-gamma (IFN-γ), and inhibit 5-lipoxygenase (5-LOX) and therefore shuts down mechanisms of leukotrienes, which are inflammatory mediators.

Many studies investigate the role of Boswellia serrata for the treatment of various inflammatory conditions of respiratory disorders such as asthma, bronchitis, and laryngitis, and cough. The anti-asthmatic potential of Boswellic acid which possesses significant anti-inflammatory activities, the data suggest that the mechanism by which it effectively treats bronchial asthma is based on reductions of Th2 cytokines via inhibition of a signal transducer and activator of transcription (pSTAT6) and GATA-3 expression and inhibit leukotriene biosynthesis which suppressed allergic airway inflammation. This treatment showed improvement of disease as evidenced by the disappearance of physical symptoms and signs such as dyspnea, rhonchi, number of attacks, as well as a decrease in the eosinophilic count.

The antiviral effect of Boswellia serrata and its components as boswellic acid was investigated against HSV-1, Chikungunya virus (CHIKV) and vesicular stomatitis virus, the mechanism of the effect of Boswellia acids against Herpes Simplex Virus (HSV) may through the inhibition of nuclear factor - kappa B (NF-κB), essential for virus replication, and observed significant down-regulation of NF-κB, and the mitogen-activated protein kinase (p38 MAP-kinase) activation, in addition, to reduce expression of tumor necrosis factor (TNF)-α, Interleukin (IL)-1β and IL-6. Also, boswellic acid had been used in the outbreak of Chikungunya virus (CHIKV) a broad antiviral agent by blocking of entry of CHIKV Env-pseudotyped lentiviral vectors and inhibited CHIKV infection in vitro.

. Pharmacokinetic studies

Aim of the work:

To evaluate the therapeutic role of Licorice extract and Boswellia serrate gum as a complementary intervention in addition to conventional therapy in Egyptian patients with COVID-19.

All included patients will be diagnosed according to the Egyptian Ministry of Health and population criteria for COVID-19 diagnosis:

Epidemiological history:

1. History of travel to or residence in communities where cases reported within 14 days prior to the onset of the disease
2. In contact with viral RNA positive people within 14 days prior to disease onset.
3. In contact with patients who have a fever or respiratory symptoms from communities confirmed cases reported within 14 days before disease onset Clinical features:

1. Fever and/or respiratory symptoms. 2. Imaging characteristics. 3. The white blood cell count was normal or decreased, with lymphocyte decreased.

Diagnosis of any suspected patient should follow the following criteria:

1. Anyone of the epidemiological history with any of the clinical features. OR
2. All three clinical features. OR
3. Severe Acute Respiratory Infection (SARI) with no other obvious cause.

Confirmed Cases:

1. RT-PCR indicates positive for novel coronavirus RNA
2. Viral specific IgM and IgG are detectable in serum
3. Viral specific IgG is detectable from negative to positive, OR
4. Viral specific IgG antibody reaches a titration of at least 4-fold higher in the recovery stage than in the acute stage.

All patients will have the following investigations:

1. X-ray chest/CT chest
2. CBC with differential count>, total blood picture
3. Arterial Blood Gas Test (ABG).
4. C-reactive protein (CRP)
5. D-Dimer.
6. Serum ferritin.
7. Triglycerides.
8. Fibrinogen.
9. Serum aspartate aminotransferase.
10. Renal functions.
11. Troponin T, Troponin I, if myocarditis is suspected. The study will be launched in at least one center related to the Ministry of Health and following the protocol recommended by the Scientific Committee and its dynamic changes that occur from time to time.

The study population will be divided into two groups of patients:

A- Group 1: Will include patients who are receiving conventional therapy according to the MOH protocol.

B- Group 2: Will include patients who will receive Licorice and Boswellia Serrata gum in addition to conventional therapy.

Dosage form:

LICORICE CAPSULES; 250 mg standardized extract (25% Glycyrrhizin - 62.5 mg).

Dose:

One capsule, Two times daily, before meals For 10 days, with measuring blood pressure daily.

Boswellia serrata Gum Resin; B. serrate contains volatile oils (5-15%), pure resin (55-66%), and mucus (12-23%). The resin contains terpenoids, phenolic compounds, flavonoids, and phenylpropanoids. More than 12 different Boswellic acids have been identified, the amounts of 11-keto-β-boswellic acid KBA is 3-4.7% and acetyl-11-keto-β-boswellic acid(AKBA) is 2.2-2.9%, Dose: 2 gm, 4 times daily For 15 days, Boswellia Gum Resin is administered by chewing for the half-hour

Statistical analysis:

All data will be analyzed statistically by using Statistical Product and Service Solutions (SPSS) version 18, to detect any statistically significant differences between the two groups which include comparing the 2 groups in all clinical and laboratory variables and statistical significance was considered when p-value <0.05, also will use univariate and multivariate analysis to show if any differences in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic and laboratory-confirmed diagnosis of COVID-19.
* RT-PCR indicates positive for novel coronavirus RNA
* Viral specific IgM and IgG are detectable in serum
* Viral specific IgG is detectable from negative to positive, OR
* Viral specific IgG antibody reaches a titration of at least 4-fold higher in the recovery stage than in the acute stage

Exclusion Criteria:

* Patients who are not fulfilling the diagnostic criteria for COVOID-19.
* Pregnant women.
* Critically ill patients who are mechanically ventilated since admission.
* Hypertensive patients.
* Congestive heart failure patients

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Increased number of people recovering from COVID-19 | 14 days
  Conversion of RT-PCR indicates positive for novel coronavirus RNA to negative

SECONDARY OUTCOMES:
Decrease number of patients that require respiratory support , | 14 days
  Decrease number of patients that require respiratory support , management in the Intensive Care Unit (ICU) and need Mechanical Ventilation Support with endotracheal intubation.
Decrease duration of hospital stay | 7 days
  Rapid recovery

CONTACTS AND LOCATIONS:
Overall Officials: Adel A. Gomaa, Ph.D., Principal Investigator — Professor of Medical pharmacology
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
A pilot study for evaluation of the potential therapeutic effect of food supplement, licorice extract, and Boswellia Serrata gum
Supporting Information: Study Protocol

REFERENCES:
- [Background] Yu X, Bao Y, Meng X, Wang S, Li T, Chang X, Xu W, Yang G, Bo T. Multi-pathway integrated adjustment mechanism of licorice flavonoids presenting anti-inflammatory activity. Oncol Lett. 2019 Nov;18(5):4956-4963. doi: 10.3892/ol.2019.10793. Epub 2019 Sep 4. PMID 31612007
- [Background] Mollica L, De Marchis F, Spitaleri A, Dallacosta C, Pennacchini D, Zamai M, Agresti A, Trisciuoglio L, Musco G, Bianchi ME. Glycyrrhizin binds to high-mobility group box 1 protein and inhibits its cytokine activities. Chem Biol. 2007 Apr;14(4):431-41. doi: 10.1016/j.chembiol.2007.03.007. PMID 17462578
- [Background] Kong D, Wang Z, Tian J, Liu T, Zhou H. Glycyrrhizin inactivates toll-like receptor (TLR) signaling pathway to reduce lipopolysaccharide-induced acute lung injury by inhibiting TLR2. J Cell Physiol. 2019 Apr;234(4):4597-4607. doi: 10.1002/jcp.27242. Epub 2018 Sep 10. PMID 30203548
- [Background] Ammon HP. Modulation of the immune system by Boswellia serrata extracts and boswellic acids. Phytomedicine. 2010 Sep;17(11):862-7. doi: 10.1016/j.phymed.2010.03.003. Epub 2010 Aug 8. PMID 20696559
- [Background] Ammon HP. Boswellic Acids and Their Role in Chronic Inflammatory Diseases. Adv Exp Med Biol. 2016;928:291-327. doi: 10.1007/978-3-319-41334-1_13. PMID 27671822
- [Background] Baram SM, Karima S, Shateri S, Tafakhori A, Fotouhi A, Lima BS, Rajaei S, Mahdavi M, Tehrani HS, Aghamollaii V, Aghamiri SH, Mansouri B, Gharahje S, Kabiri S, Hosseinizadeh M, Shahamati SZ, Alborzi AT. Functional improvement and immune-inflammatory cytokines profile of ischaemic stroke patients after treatment with boswellic acids: a randomized, double-blind, placebo-controlled, pilot trial. Inflammopharmacology. 2019 Dec;27(6):1101-1112. doi: 10.1007/s10787-019-00627-z. Epub 2019 Aug 12. PMID 31407195
- [Background] Beghelli D, Isani G, Roncada P, Andreani G, Bistoni O, Bertocchi M, Lupidi G, Alunno A. Antioxidant and Ex Vivo Immune System Regulatory Properties of Boswellia serrata Extracts. Oxid Med Cell Longev. 2017;2017:7468064. doi: 10.1155/2017/7468064. Epub 2017 Mar 13. PMID 28386311
- [Background] Eltahir HM, Fawzy MA, Mohamed EM, Alrehany MA, Shehata AM, Abouzied MM. Antioxidant, anti-inflammatory and anti-fibrotic effects of Boswellia serrate gum resin in CCl4-induced hepatotoxicity. Exp Ther Med. 2020 Feb;19(2):1313-1321. doi: 10.3892/etm.2019.8353. Epub 2019 Dec 19. PMID 32010304
- [Background] Goswami D, Mahapatra AD, Banerjee S, Kar A, Ojha D, Mukherjee PK, Chattopadhyay D. Boswellia serrata oleo-gum-resin and beta-boswellic acid inhibits HSV-1 infection in vitro through modulation of NF-small ka, CyrillicB and p38 MAP kinase signaling. Phytomedicine. 2018 Dec 1;51:94-103. doi: 10.1016/j.phymed.2018.10.016. Epub 2018 Oct 16. PMID 30466633
- [Background] Zhou X, Cai JG, Zhu WW, Zhao HY, Wang K, Zhang XF. Boswellic acid attenuates asthma phenotype by downregulation of GATA3 via nhibition of PSTAT6. Genet Mol Res. 2015 Jul 6;14(3):7463-8. doi: 10.4238/2015.July.3.22. PMID 26214425
- [Background] Loeser K, Seemann S, Konig S, Lenhardt I, Abdel-Tawab M, Koeberle A, Werz O, Lupp A. Protective Effect of Casperome(R), an Orally Bioavailable Frankincense Extract, on Lipopolysaccharide- Induced Systemic Inflammation in Mice. Front Pharmacol. 2018 Apr 20;9:387. doi: 10.3389/fphar.2018.00387. eCollection 2018. PMID 29731716
- [Background] Roy NK, Parama D, Banik K, Bordoloi D, Devi AK, Thakur KK, Padmavathi G, Shakibaei M, Fan L, Sethi G, Kunnumakkara AB. An Update on Pharmacological Potential of Boswellic Acids against Chronic Diseases. Int J Mol Sci. 2019 Aug 22;20(17):4101. doi: 10.3390/ijms20174101. PMID 31443458
- [Background] Soni KK, Meshram D, Lawal TO, Patel U, Mahady GB. Fractions of Boswellia Serrata Suppress LTA4, LTC4, Cyclooxygenase-2 Activities and mRNA in HL-60 Cells and Reduce Lung Inflammation in BALB/c Mice. Curr Drug Discov Technol. 2021;18(1):95-104. doi: 10.2174/1570163817666200127112928. PMID 31985381
- [Background] von Rhein C, Weidner T, Henss L, Martin J, Weber C, Sliva K, Schnierle BS. Curcumin and Boswellia serrata gum resin extract inhibit chikungunya and vesicular stomatitis virus infections in vitro. Antiviral Res. 2016 Jan;125:51-7. doi: 10.1016/j.antiviral.2015.11.007. Epub 2015 Dec 2. PMID 26611396
- [Background] Cinatl J, Morgenstern B, Bauer G, Chandra P, Rabenau H, Doerr HW. Glycyrrhizin, an active component of liquorice roots, and replication of SARS-associated coronavirus. Lancet. 2003 Jun 14;361(9374):2045-6. doi: 10.1016/s0140-6736(03)13615-x. PMID 12814717
- [Background] Redeploying plant defences. Nat Plants. 2020 Mar;6(3):177. doi: 10.1038/s41477-020-0628-0. PMID 32170291
- [Background] Wang L, Yang R, Yuan B, Liu Y, Liu C. The antiviral and antimicrobial activities of licorice, a widely-used Chinese herb. Acta Pharm Sin B. 2015 Jul;5(4):310-5. doi: 10.1016/j.apsb.2015.05.005. Epub 2015 Jun 17. PMID 26579460
- [Background] Sun ZG, Zhao TT, Lu N, Yang YA, Zhu HL. Research Progress of Glycyrrhizic Acid on Antiviral Activity. Mini Rev Med Chem. 2019;19(10):826-832. doi: 10.2174/1389557519666190119111125. PMID 30659537
- [Background] Luo P, Liu D, Li J. Pharmacological perspective: glycyrrhizin may be an efficacious therapeutic agent for COVID-19. Int J Antimicrob Agents. 2020 Jun;55(6):105995. doi: 10.1016/j.ijantimicag.2020.105995. Epub 2020 Apr 24. PMID 32335281
- [Background] Guo A, He D, Xu HB, Geng CA, Zhao J. Promotion of regulatory T cell induction by immunomodulatory herbal medicine licorice and its two constituents. Sci Rep. 2015 Sep 15;5:14046. doi: 10.1038/srep14046. PMID 26370586
- [Background] Li X, He X, Liu B, Xu L, Lu C, Zhao H, Niu X, Chen S, Lu A. Maturation of murine bone marrow-derived dendritic cells induced by Radix Glycyrrhizae polysaccharide. Molecules. 2012 May 30;17(6):6557-68. doi: 10.3390/molecules17066557. PMID 22728353
- [Derived] Gomaa AA, Mohamed HS, Abd-Ellatief RB, Gomaa MA, Hammam DS. Advancing combination treatment with glycyrrhizin and boswellic acids for hospitalized patients with moderate COVID-19 infection: a randomized clinical trial. Inflammopharmacology. 2022 Apr;30(2):477-486. doi: 10.1007/s10787-022-00939-7. Epub 2022 Mar 1. PMID 35233748
- [Derived] Armanini D, Fiore C, Bielenberg J, Sabbadin C, Bordin L. Coronavirus-19: Possible Therapeutic Implications of Spironolactone and Dry Extract of Glycyrrhiza glabra L. (Licorice). Front Pharmacol. 2020 Oct 22;11:558418. doi: 10.3389/fphar.2020.558418. eCollection 2020. PMID 33192504